CLINICAL TRIAL: NCT05601466
Title: Clinical Study on QN-023a Targeting CD33 in Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: Natural Killer(NK) Cell Therapy for Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: It did not reach the expected results of clinical trial
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: Hangzhou Qihan Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2022029
Record Dates: First submitted 2022-10-21; First posted 2022-11-01 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-05

CONDITIONS: AML, Adult
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cyclophosphamide; fludarabine; Cytarabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QN-023a (Experimental): QN-023a in adult subjects with r/r AML
  Interventions: Drug: QN-023a; Drug: Cyclophosphamid; Drug: Fludarabine; Drug: Cytarabine

INTERVENTIONS:
Drug: QN-023a — NK cell therapy
Drug: Cyclophosphamid — Lympho-conditioning Agent
Drug: Fludarabine — Lympho-conditioning Agent
Drug: Cytarabine — Lympho-conditioning Agent

SUMMARY:
This is an open-label, Phase I study of QN-023a (allogeneic CAR-NK cells targeting CD33) in relapsed/refractory Acute Myeloid Leukemia (AML).

The clinical study is to evaluate the safety, tolerability and preliminary efficacy of QN-023a in patients with relapsed/refractory AML,where a "3+3" enrollment schema will be utilized at dose escalation stage. Up to 18 patients will be enrolled.

ELIGIBILITY:
Key Inclusion Criteria:

* Provision of signed and dated informed consent form (ICF)
* ≥18 years old
* Diagnosis of r/r AML
* Subjects with CD33 positive leukemia cells
* Eastern Cooperative Oncology Group (ECOG) performance status ≤1
* Adequate organ function as defined in the protocol
* Donor specific antibody (DSA) to QN-023a: MFI <= 2000

Key Exclusion Criteria:

* Allergic to drug used in this study
* Accept other anti-tumor drug within certain time of day 0 (first QN-023a dose infusion), time window and drug defined in the protocol.
* received systemic immunosuppressive therapy within 7 days of day 0, or likely to require systemic immunosuppressive therapy
* Acute Promyelocytic Leukemia (APL)
* Active central nervous system Leukemia.
* Uncontrolled, active clinically significant infection
* Clinically significant cardiovascular disease as defined in the protocol
* Known HIV infection, active Hepatitis B (HBV) or Hepatitis C (HCV) infection
* History of central nervous system (CNS) disease such as stroke, epilepsy.
* Females are pregnant or lactating
* Investigator-assessed presence of any medical or social issues that are likely to interfere with study conduct or may cause increased risk to subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2022-03-26 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-11 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 28 Days from first dose of QN-023a
The incidence of subjects with Dose Limiting Toxicities within each dose level cohort | 28 Days from first dose of QN-023a

SECONDARY OUTCOMES:
Overall Response Rate(ORR) | Up to approximately 2 years after last dose of QN-023a
Relapse-free survival (RFS) of participants | Up to approximately 2 years after last dose of QN-023a
Determination of the pharmacokinetics (PK) of QN-023a cells in peripheral blood | Up to approximately 2 years after last dose of QN-023a
  The PK of QN-023a in peripheral blood will be reported as the relative percentage of product (QN-023a) DNA versus patient DNA (% chimerism) measured from blood samples at the specified time points

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No